CLINICAL TRIAL: NCT04486248
Title: Comparison of Magnetic Resonance Techniques for the Measurement of Cerebral Blood Perfusion
Status: Completed | Type: Observational
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ASL/BBRC2019
Record Dates: First submitted 2020-07-20; First posted 2020-07-24 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2021-09

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this project, we aim at implementing a te-ASL sequence and to compare it to two reference ASL sequences with a fixed PLD on healthy individuals. On the one hand, the te-ASL sequence will be compared against a 3D pCASL with a PLD of 1800 ms, as the current reference according the Consensus of the ISMRM perfusion study group and the European consortium for ASL in dementia. On the other, as the implemented te-ASL sequence will have a 2D readout, it will also be compared to a 2D pCASL ASL sequence with the same PLD, in order to be able to disentangle differences due to the dynamic PLD scheme from those arising from the different read-out schemes.

ELIGIBILITY:
Inclusion Criteria:

* To sign the study informed consent form approved by the corresponding authorities.
* Healthy men and women (older than 18 years old).

Exclusion Criteria:

* Inability or unwillingness to give written informed consent or communicate with the study staff or illiteracy.
* Any contraindication to perform brain MRI procedure (e.g. pacemaker, MRI-incompatible aneurysm clips).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty (N=30) healthy individuals older than 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
ASL perfusion MRI data | Through study completion, an average of 1 year
  Quantification of cerebral blood flow

CONTACTS AND LOCATIONS:
Locations (1):
- BarcelonaBeta Brain Research Center, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided